CLINICAL TRIAL: NCT03934671
Title: Evaluation of the Efficacy of an Antioxidant Dressing in Chronic Wound Healing
Acronym: REOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: Histocell, S.L. (Industry); Andalusian Health Service: District Poniente Almería. (Unknown); Andalusian Health Service: District Jaén (Unknown); Andalusian Health Service: District Jaén-Nordeste (Unknown); Andalusian Health Service: Health Management Area Este of Málaga-Axarquía. (Unknown)
Responsible Party: Principal Investigator, Inés María Comino-Sanz, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TD-REOX-2019
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Hard-to-heal Wounds
Keywords: Chronic wound; Wound healing; Hard-to-heal wounds; Antioxidant dressing; Oxidative stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant dressing (active product) (Experimental)
  Interventions: Device: Antioxidant dressing (active product)
- Usual care dressing (standard clinical practice) (Active Comparator)
  Interventions: Device: Usual care dressing that create a moist environment (standard clinical practice)

INTERVENTIONS:
Device: Antioxidant dressing (active product) — Antioxidant dressing (active product), covered with secondary dressing. Compression bandage if necessary.
  Device: Reoxcare®
  Arms: Antioxidant dressing (active product)
Device: Usual care dressing that create a moist environment (standard clinical practice) — Usual care dressing; moist environment dressing chosen from the study centres' formulary (hydrocolloid, alginate, polyurethane foam dressings, silver dressings). Compression bandage if necessary
  Arms: Usual care dressing (standard clinical practice)

SUMMARY:
The aim of this study is to compare the effect of antioxidant dressing (active product) on chronic wound healing with the use of non-active wound dressing for healing in a moist environment (standard clinical practice) in patients with hard-to-heal wounds

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with leg ulcers (venous, ischemic, traumatic or diabetic foot ulcer).
* Patients with dehisced surgical wounds healing by second intention.
* Patients with pressure ulcers.
* Wound area between 1 and 250 cm2.

Exclusion Criteria:

* Systemic inflammatory disease or oncological disease.
* Wounds with clinical signs of infection.
* Terminal situation (life expectancy less than 6 months).
* Ulcers from other etiologies: tumours, infectious.
* Wounds treated with negative pressure therapy.
* Pregnancy.
* History of sensitivity or allergy to any of the components of the study dressing.

In addition, criteria for withdrawal from the study will be considered:

* Worsening of the wound according to the clinical judgment of the professional (appearance of clinical signs of infection or others).
* Appearance of allergies or hypersensitivity to the dressing.
* Death.
* Hospital admission that interrupts or complicates the continuity of care in the Nursing Consultation.
* Transfer to another Health District where there can be no continuity of care with the active dressing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the score of the RESVECH 2.0 scale for chronic wound healing monitoring | At baseline, after 2 week, after 4 week, after 6 week and after 8 week
  The RESVECH 2.0 is a scale for monitoring the cicatrization of the wound. It has 6 items: size of the lesion, depth/tissue concerned, edges, type of tissue in the wound bed, exudate, infection/inflammation. The scale is scored numerically and can score ranging from 0 to 35 points, wound healed and the worst possible lesion respectively
Wound size reduction | At baseline, after 2 week, after 4 week, after 6 week and after 8 week
  Difference in wound area between first and last dressing

SECONDARY OUTCOMES:
Time required to achieve 50% reduction in wound size | Change from baseline to 8 weeks of follow up
Time to removal of non-viable tissue from wound bed | At baseline, after 2 week, after 4 week, after 6 week and after 8 week
Number of completely healed wounds | At baseline, after 2 week, after 4 week, after 6 week and after 8 week
Pain level | At baseline, after 2 week, after 4 week, after 6 week and after 8 week
  The visual analogue scale (VAS) is commonly used as the outcome measure for patient´s pain. It is usually presented as a 100-mm horizontal line on which pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Area of wound with bacterial load | At baseline, after 2 week, after 4 week, after 6 week and after 8 week
  clinical signs of infection and/or measurement of surfaces with bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Jaén, Jaén, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Castro B, Bastida FD, Segovia T, Lopez Casanova P, Soldevilla JJ, Verdu-Soriano J. The use of an antioxidant dressing on hard-to-heal wounds: a multicentre, prospective case series. J Wound Care. 2017 Dec 2;26(12):742-750. doi: 10.12968/jowc.2017.26.12.742. PMID 29244974
- [Background] Castro B, Palomares T, Azcoitia I, Bastida F, del Olmo M, Soldevilla JJ, Alonso-Varona A. Development and preclinical evaluation of a new galactomannan-based dressing with antioxidant properties for wound healing. Histol Histopathol. 2015 Dec;30(12):1499-512. doi: 10.14670/HH-11-646. Epub 2015 Jul 3. PMID 26140672
- [Background] Comino-Sanz IM, Lopez-Franco MD, Castro B, Pancorbo-Hidalgo PL. Antioxidant dressing therapy versus standard wound care in chronic wounds (the REOX study): study protocol for a randomized controlled trial. Trials. 2020 Jun 8;21(1):505. doi: 10.1186/s13063-020-04445-5. PMID 32513260
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29244974
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/26140672